CLINICAL TRIAL: NCT00973557
Title: The Effect of Monoclonal Vascular Endothelial Growth Factor (VEGF) Antibody (Bevacizumab) on Pituitary Function
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, William Gellepis, Research Administrator, Cedars-Sinai Medical Center
Other Study IDs: Pro00019830
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer; Lung Cancer; Breast Cancer; Glioblastoma
Keywords: bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 10 ml of whole blood will be collected to measure prolactin, growth hormone, IGF-I, TSH, thyroxine, ACTH, and cortisol levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Taking Bevacizumab: Patients who are currently being treated for cancer by the drug Bevacizumab.

SUMMARY:
The purpose of this research is to determine whether the drug, Bevacizumab (a monoclonal anti VEGF-A antibody), which is approved to treat patients with metastatic colon cancer induces hyperprolactinemia (increased prolactin secretion) in humans with intact pituitary function. Past studies have shown Bevacizumab to shrink tumor size and also increase prolactin levels. The mechanism of the hyperprolactinemia might be inhibition of pituitary portal vein transport, suggesting that Bevacizumab induces prolactin secretion from normal lactotrophs in the pituitary gland.

Patients who have been treated with Bevacizumab for at least one month will be recruited to participate.

The subjects who are being treated with Bevacizumab by Dr. Stephen Wolin (a sub-investigator) will be screened by him for study eligibility. Dr. Wolin will approach eligible patients with all the information and background of the study and see if they have an interest in being consented.

If consented, there will be 2 blood draws for the research that is not part of their standard care in which 10 ml of blood is collected and prolactin, growth hormone, IGF-I, TSH, thyroxine, ACTH, and cortisol will be measured. One 5ml blood draw will occur before the administration of Bevacizumab and the second 5 ml blood draw will occur after the administration of the Bevacizumab. The investigators will then review the laboratory results. The blood tests are of the hormones of the pituitary gland to test pituitary function and see if there are any abnormalities with the secretions of the gland. Pituitary function abnormalities and hyperprolactinemia are diagnosed by looking at hormone levels in the blood and comparing them to the normal reference ranges.

This study will only involve 10 subjects and will be conducted entirely at Cedars-Sinai Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer, lung cancer, breast cancer, and glioblastoma patients that have been treated with Bevacizumab for at least 1 month
* Adults (18 years of age or older)

Exclusion Criteria:

* Patients who are taking medications known to affect serum prolactin levels
* Patients who are pregnant
* Patients who have pituitary disease
* Minors (Under the age of 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have cancer and have been treated with the drug Bevacizumab for at least one month.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine whether the drug, Bevacizumab (a monoclonal anti VEGF-A antibody), which is approved to treat patients with metastatic colon cancer induces hyperprolactinemia (increased prolactin secretion) in humans with intact pituitary function. | 6 weeks
  Patients will have their blood drawn before their first Bevacizumab infusion and then again 6 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Korsisaari N, Ross J, Wu X, Kowanetz M, Pal N, Hall L, Eastham-Anderson J, Forrest WF, Van Bruggen N, Peale FV, Ferrara N. Blocking vascular endothelial growth factor-A inhibits the growth of pituitary adenomas and lowers serum prolactin level in a mouse model of multiple endocrine neoplasia type 1. Clin Cancer Res. 2008 Jan 1;14(1):249-58. doi: 10.1158/1078-0432.CCR-07-1552. PMID 18172277